CLINICAL TRIAL: NCT04080973
Title: Metabolic Workup in Patients Suffering From Kidney Stone Disease and Show Osteopenic Bone Changes on Non-contrast CT Scan
Brief Title: Metabolic Workup in Patients Suffering From Kidney Stone Disease and Osteopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0141-18-ZIV
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Urolithiasis; Renal Colic; Osteopenia
Keywords: urolithiasis; metabolic abnormalities; osteopenia; hypercalcemia; hypercalcuria; bone density
MeSH Terms: conditions — Urolithiasis; Renal Colic; Bone Diseases, Metabolic; Hypercalcemia; Hypercalciuria | interventions — Tomography, X-Ray Computed; Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: cohort study of all patients presenting with renal colic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osteopenic patients (Experimental): patients with a kidney stone and osteopenic changes.
  Interventions: Diagnostic Test: CT scan; Diagnostic Test: 24 hour urine collection

INTERVENTIONS:
Diagnostic Test: CT scan — non contrast spiral CT of the urinary tract including the bony structures of the spine and pelvis
Diagnostic Test: 24 hour urine collection — 24 hours collection of urine and measurement of the concentration of calcium, phosphorous, uric acid, oxalate and citrate
  Other Names: uninalysis

SUMMARY:
Patients suffering from acute renal colic are evaluated by non contrast computerized tomography with excellent identification rates of urinary stones. The scan also covers the bones of the ribs, spine and pelvis, allowing measurements of the bone density and identifying early osteopenic changes. Bone demineralization is associated with metabolic changes such as hypercalcemia or hypercalcuria. In this study the investigators will look for correlation between kidney stones, osteopenic bone changes and metabolic abnormalities.

DETAILED DESCRIPTION:
Kidney stones are a common medical condition found in more then 5% of the adult population. The stones might cause severe pain (due to acute obstruction of a renal unit) , deterioration of renal function and urinary tract infection. One of the causes of kidney stones is metabolic changes such as hypercalcemia or hyperoxaluria. Basic evaluation of kidney stones patients include measurements of calcium, phosphor and uric acid in the serum and is often negative. Thorough metabolic workup including 24 hours urine collection is not cost effective and is reserved for patients with frequent recurrence of stone disease.

Metabolic abnormalities are often associated with bone demineralization, of which the patients are typically unaware. such changes can be detected by the CT scan. On the same scan, performed for identifying the stone, the radiologist can measure bone density, using the Hounsfield units, in the L2 vertebral body of and the acetabular area of the pelvis.

In the study, in all patients undergoing CT scan due to renal colic, the bone density will be measured. Patients with abnormal bone density will undergo a complete metabolic workup including 24 hours collection of urine and measurements of urinary clearance of calcium, phosphorous, uric acid, oxalate and citrate . The investigators will look for correlation between osteopenic changes and metabolic abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or old
* informed consent
* kidney stones
* CT scan positive for stones AND bone changes

Exclusion Criteria:

* under 18
* unable to sign
* no stones detected on scan (even if a stone was expelled recently)
* no bone changes
* pregnancy
* a patient already known to suffer from metabolic bone disease
* a patient with documented osteoporosis
* patients following spinal or pelvic trauma / surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
correlation between abnormal metabolic changes and abnormal bone density on Ct scan | 1 year
  The rate of patients presenting with kidney stones and abnormal bone density and have abnormal urinary clearance of electrolytes.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Katz, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ran Katz, Safed, Israel

IPD SHARING:
Plan to Share IPD: No